CLINICAL TRIAL: NCT00002043
Title: Dapsone 100 Mg Versus 50 as Primary Prophylaxis for Pneumocystis Carinii Pneumonia (PCP) in Patients With AIDS-Related Complex (ARC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobus Pharmaceutical (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 007B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-12

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Leukoplakia, Oral; Dapsone; AIDS-Related Complex; Candidiasis, Oral
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Leukoplakia, Oral; AIDS-Related Complex; Candidiasis, Oral | interventions — Dapsone

INTERVENTIONS:
Drug: Dapsone

SUMMARY:
To determine which of 2 doses of dapsone is effective prophylaxis for Pneumocystis carinii pneumonia (PCP) in patients with oral thrush or hairy leukoplakia and less than 400 CD4 lymphocytes per mm3. To determine whether the long-term toxicities associated with daily dapsone in this population are tolerable.

ELIGIBILITY:
Inclusion Criteria

The patient must have HIV positive antibody test and presence of oral thrush or hairy leukoplakia.

* Patient must be willing and able to sign informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Prior Pneumocystis carinii pneumonia (PCP) or AIDS-defining condition.
* Prophylaxis for PCP in preceding 3 months.
* Absence of detectable glucose-6-phosphate dehydrogenase (G6PD) activity.
* Prior type I hypersensitivity (anaphylaxis, urticaria, angioedema) or exfoliative dermatitis during treatment with dapsone.
* History of poor compliance.

Concurrent Medication:

Excluded:

* Zidovudine (AZT).

Patients with the following are excluded:

* Prior Pneumocystis carinii pneumonia (PCP) or AIDS-defining condition.
* Prophylaxis for PCP in preceding 3 months.
* Absence of detectable glucose-6-phosphate dehydrogenase (G6PD) activity.
* Concurrent or prior therapy with zidovudine (AZT).
* Prior type I hypersensitivity (anaphylaxis, urticaria, angioedema) or exfoliative dermatitis during treatment with dapsone.
* History of poor compliance.

Prior Medication:

Excluded:

* Zidovudine (AZT).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA CARE Ctr, Los Angeles, California, United States